CLINICAL TRIAL: NCT06254131
Title: Preoperative Ondansetron Lozenge for Prevention of Postoperative Nausea and Vomiting in Caesarean Section: A Randomized Controlled Trial
Brief Title: Preoperative Ondansetron Lozenge for Prevention of Postoperative Nausea and Vomiting in Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ِAhmed Mohamed Ibrahim, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264PR460/12/2023
Record Dates: First submitted 2024-01-27; First posted 2024-02-12 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Ondansetron Lozenge; Postoperative Nausea and Vomiting; Caesarean Section
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ondansetron lozenge (Ondalenz ©) (Experimental): Patients will receive ondansetron lozenge 4 mg (Ondalenz ©), 2 hours before surgery.
  Interventions: Drug: Ondansetron lozenge (Ondalenz ©)
- Ondansetron IV (Experimental): Patients will receive 4 mg of ondansetron IV approximately 30 minutes before the end of surgery.
  Interventions: Drug: Ondansetron IV
- Control group (No Intervention): Patients will not receive ondansetron as a control group.

INTERVENTIONS:
Drug: Ondansetron lozenge (Ondalenz ©) — Patients will receive ondansetron lozenge 4 mg (Ondalenz ©), 2 hours before surgery.
  Arms: Ondansetron lozenge (Ondalenz ©)
Drug: Ondansetron IV — Patients will receive 4 mg of ondansetron IV approximately 30 minutes before the end of surgery.
  Arms: Ondansetron IV

SUMMARY:
The aim of this study is to estimate the effect of preoperative ondansetron lozenge on prevention of postoperative nausea and vomiting in caesarean section.

DETAILED DESCRIPTION:
Caesarean section has become increasingly popular, and it is the most performed surgical procedure. Despite consciousness allowing the patient to have an early intimate bond with the newborn, the procedure may be associated with complications. Around 30% of individuals undergoing elective procedures under general anesthetic are affected by postoperative nausea and vomiting (PONV).

PONV may decrease the quality of recovery and cause aspiration, intracranial hypertension, dehydration, acid-base disturbance, electrolyte imbalance, and neurological deterioration which leads to a prolonged hospital stay and increased medical cost.

The latest guidelines for the management of PONV recommend the administration of prophylactic antiemetic drugs (AED) as part of a multimodal therapy in high-risk adults.

Ondansetron is generally considered to be the first-line antiemetic for patients because of its favorable side effect profile. Ondansetron reduces the activity of the vagus nerve, which deactivates the vomiting center in the medulla oblongata, and also blocks serotonin receptors in the chemoreceptor trigger zone, Ondansetron is an effective drug in the prevention and treatment of PONV by having low side effects

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 35 years old.
* American Society of Anesthesiologists (ASA) physical status II.
* Undergoing caesarean section under general anesthesia.

Exclusion Criteria:

* Medical history of alcohol or drug abuse.
* History of allergic reactions or intolerance to any study medications.
* BMI > 40 kg/m2.
* History of nausea and/or vomiting within 24 h prior procedures.
* History of treatment with antiemetic medication for nausea or vomiting within 24 h of their procedure.
* History of chemotherapy treatment within 4 weeks prior to surgery.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women caesarean section
Enrollment: 75 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) | 24 hours postoperatively
  The incidence of nausea and vomiting will be evaluated through the Bellville scoring scale (lack of nausea and vomiting=0, nausea=1, nausea with belching=2, and vomiting=3).

SECONDARY OUTCOMES:
Severity of postoperative nausea and vomiting (PONV) | 24 hours postoperatively
  Severity of postoperative nausea and vomiting will be scored at 0-4, 4-12, 12-24 hours using Nausea vomiting scores (NVS): [(0, No complaint; 1, Mild degree of nausea; 2, Moderate degree of nausea; 3, Frequent vomiting; 4, Severe vomiting (continuously)].
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale Patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied ; 5, extremely satisfied).
Adverse effects | 24 hours postoperatively
  Side effects including headache, dry mouth, dizziness, visual disturbances, agitation, and sedation, will be evaluated on admission to the post anesthesia care unit (PACU) until discharge from the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.